CLINICAL TRIAL: NCT03077399
Title: Clinical Validation of SCALA, a New Rating Scale for Assessing Lateropulsion After Stroke
Brief Title: Validation Study of SCALA, Scale for Lateropulsion
Acronym: SCALA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC16.088
Record Dates: First submitted 2016-10-07; First posted 2017-03-13 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Stroke
Keywords: lateropulsion; stroke; Pusher syndrome
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: This study is a monocentric observational clinical study. During the first week, the assessments used in routine in our center will be performed. During the second week, the assessments of lateropulsion by SCALA-V1, postural verticality perception in sitting and the representation of longitudinal body axis in lying position will be performed twice, 2 days apart, by 2 different raters in order to determine their inter-rater reliability. During the third week, mass distribution on lower limbs in frontal plan during standing position and body orientation in frontal plan during sitting position, standing position and sit-to-stand will be assessed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stroke (Experimental): stroke patients, application of SCALA
  Interventions: Device: SCALA
- control (Experimental): Healthy individuals (patients without stroke), application of SCALA
  Interventions: Device: SCALA

INTERVENTIONS:
Device: SCALA — All items of SCALA are applied

SUMMARY:
Development and clinical validation of SCALA, a new rating scale for lateropulsion after stroke. A monocentric clinical study including 78 post-stroke individuals and 30 patients without stroke and/or healthy volunteers.

In order to analyze the SCALA's content validity, a Delphi-type consensus process was applied prior to clinical validation. The Delphi process, including 20 international experts, has given rise to the version of the scale to be tested clinically (SCALA-V1; Paper in preparation).

DETAILED DESCRIPTION:
The protocol aims to develop and validate a new clinical rating scale assessing lateropulsion after stroke. The project is driven by the need to have a tool that better meets clinometric properties than the 2 main existing scales, the Scale for Contraversive Pushing (SCP) and the Burke Lateropulsion Scale (BLS), and by the need to have a unicist scale to assess all components of lateropulsion (i.e. body tilt, active pushing by non-paretic limbs and resistance to passive correction) regardless the mechanisms or the severity of lateropulsion and the side of the stroke lesion.

The initial version (version 0) of the scale has been developed by our team in Grenoble (SCALA-V0). In a first step, an online expert consensus process (Delphi method) will give rise to a version 1 (SCALA-V1), considered as generally accepted by the scientific community.

The SCALA-V1 will be validated in a monocentric clinical study. 78 individuals with stroke and 30 individuals without stroke and/or healthy controls will be included.

All subjects will be comprehensively assessed during 3 weeks. During the first week will be performed many assessments used in routine in our center. These assessments will serve to describe participants and ensure that our series is comparable to others of the literature. These assessments which are not considered as outcome are: age, sex, height, weight, manual laterality, comorbidity, apraxia, executive function deficits, retropulsion, depression, and autonomy. Several other clinical assessments will also be performed during the first week, this time to serve as outcomes: stroke lesion characteristics, motor weakness, spasticity, spatial neglect, anosognosia, aphasia, hemianopsia, hypoesthesia, visual verticality, balance and gait disorders. During the second week, lateropulsion by SCALA-V1, verticality perception and spatial representation will be assessed to determine their inter-rater reliability. During the last week, mass distribution on lower limbs in frontal plan during standing position and body orientation in frontal plan during sitting position, standing position and sit-to-stand will be assessed.

Editorial valorization of the clinical trial: This study will be valorized by several papers, one concerning clinometric properties of SCALA-V1 (reliability …), other(s) paper(s) about the understanding of lateropulsion, and clinometric properties of the devices assessing vertical perception and body orientation.

ELIGIBILITY:
Inclusion Criteria: All types of stroke, ≤6 months.

Exclusion Criteria: postural disorders other than stroke or body geometry disorders (e.g. limb amputation, severe deformity, bone fracture, trunk deformity with deviation of C7 greater than 30mm) interfering with balance, acute vertigo, history of severe psychiatric disease, medical instability, dementia diagnosed, and severe understanding deficits limiting assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
SCALA Reliability | week 2 (assessed twice +/-2d)
  Inter-rater reliability, internal consistency, measurement error of SCALA

SECONDARY OUTCOMES:
Influence of vision on lateropulsion | week 2
  Comparison of scores of items performed with and without vision
Interest of the condition without vision on the lateropulsion diagnosis from the SCALA total score. | week 2
  Comparison of proportion of individuals with a lateropulsion by using the total score of SCALA based on all items (with and without vision) and that of individuals with a lateropulsion by using the total score of SCALA based only on items with vision
Evaluation of SCALA feasibility | Week 2
  Influence of sensory-motor, language and cognitive deficits, severity of balance and gait disorders, and stroke features (type and localization) on the time required to complete SCALA; Descriptive statistics on items judged as "not applicable"
To improve the understanding of mechanisms underpinning lateropulsion | weeks 1,2 and 3
  Relation between the total score or subscores of SCALA, and stroke lesion characteristics, verticality perception, representation of longitudinal body axis in lying position, body orientation in frontal plan, weight-bearing asymmetry, and awareness of deficits.
Reliability of supplementary instrumental assessments of lateropulsion | Week 2 (assessed twice +/-2d)
  Inter-rater reliability of longitudinal body axis representation and postural verticality perception
Criterion validity of SCALA | Weeks 1 and 2
  Comparison to Scale for Contraversive Pushing and Burke Lateropulsion Scale, which currently are considered as gold-standards to assess lateropulsion.
Descriptive analysis of data of individuals with stroke | Weeks 1, 2 and 3
  Descriptive analysis of data
Descriptive analysis of data of healthy controls | Day 1
  Descriptive analysis of data including normality ranges.

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Pérennou, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital, Grenoble, France

IPD SHARING:
Plan to Share IPD: No